CLINICAL TRIAL: NCT05434091
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO CONTROLLED, 4-PERIOD, CROSSOVER, FIRST-IN-HUMAN STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF SINGLE ASCENDING ORAL DOSES OF PF 07291177 ADMINISTERED TO HEALTHY ADULT PARTICIPANTS
Brief Title: A First-In-Human Study of the Study Medicine, Called PF-07291177, in Healthy Adult Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopped due to change in strategy.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: C4741003; 2022-500253-17-00 (Other: EU CTIS)
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Healthy Participants
Keywords: PF-07291177; Single ascending dose; Transthyretin; Retinol binding protein; Healthy participants; Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- PF-07291177 and Placebo (Cohort 1) (Experimental): Single dose administration of PF-07291177 and placebo; Within a cohort, participants will receive 3 doses of PF-07291177 and 1 dose of placebo.
  Interventions: Drug: PF-07291177; Drug: Placebo
- PF-07291177 and Placebo (Cohort 2) (Experimental): Single dose administration of PF-07291177 and placebo; Within a cohort, participants will receive 3 doses of PF-07291177 and 1 dose of placebo.
  Interventions: Drug: PF-07291177; Drug: Placebo
- PF-07291177 and Placebo (Cohort 3) (Experimental): Single dose administration of PF-07291177 and placebo; Within a cohort, participants will receive 3 doses of PF-07291177 and 1 dose of placebo.
  Interventions: Drug: PF-07291177; Drug: Placebo

INTERVENTIONS:
Drug: PF-07291177 — PF-07291177 will be prepared as an oral solution and/or suspension given in escalating single doses to be determined
Drug: Placebo — Matching placebo will be prepared as an oral solution and/or suspension given in each cohort

SUMMARY:
The purpose of the study is to learn about the safety, tolerability (the extent to which side effects can be tolerated), and plasma pharmacokinetics (PK) (PK helps us understand how the drug is changed and eliminated from body after you take it) of PF-07291177 after administration of escalating, single, doses by mouth.

DETAILED DESCRIPTION:
The purpose of the study is to learn about the safety, the extent to which side effects can be tolerated, and plasma pharmacokinetics (PK) (PK helps us understand how the drug is changed and eliminated from your body after you take it) of PF-07291177 after administration of escalating, single, doses by mouth.

Each participant in this study is planned to undergo up to 4 treatment periods receiving up to 3 doses of PF 07291177 and 1 dose of placebo.

Precautionary sentinel dosing will be used in this study. Two participants (1 receiving PF 07291177 and 1 receiving placebo) within a period will be dosed initially before the remaining participants of that period are dosed.

This study is seeking :

* Female participants of non-child bearing potential and males must be 18 to 60 years of age, inclusive, at the time of signing the ICD
* Female participants of non-child bearing potential and males who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.

ELIGIBILITY:
This study is seeking participants who are:

1. Female participants of non-child bearing potential and males must be 18 to 60 years of age, inclusive, at the time of signing the inform consent documents.
2. Female participants of non-child bearing potential and males who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

This study is not seeking participants who have:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to coronavirus disease 2019 (COVID-19) pandemic that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
3. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention, with the exception of moderate/strong cytochrome P450 3A inducers or time-dependent inhibitors which are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention.
4. Received a COVID-19 vaccine within 7 days before screening or any visit in which a safety lab is planned, or who are to be vaccinated with a COVID-19 vaccine within 7 days before screening or any visit in which a safety lab is planned.
5. Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
6. Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest.
7. Renal impairment as defined by an estimated glomerular filtration rate (eGFR) <75 mL/min/1.73m2
8. Standard 12 lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete left bundle branch block (LBBB), signs of an acute or indeterminate age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the uncorrected QT interval is >450 ms, this interval should be rate corrected using the Fridericia method only and the resulting QTcF should be used for decision making and reporting.
9. ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

   * Aspartate aminotransferase or Alanine aminotransferase level ≥1.25× upper limit of normal (ULN);
   * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.
10. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit, or 3 ounces (90 mL) of wine).
11. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2023-03-29 (Estimated); Study Completion 2023-03-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline up to 35 days after last dose of study intervention (approximately 11 weeks)
Number of Participants With Clinical Laboratory Abnormalities | Baseline up to 10 days after last dose of study intervention (approximately 5 weeks)
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to 10 days after last dose of study intervention (approximately 5 weeks)
Number of Participants With Change From Baseline in Electrocardiogram (ECG) Findings | Baseline up to 10 days after last dose of study intervention (approximately 5 weeks)
Number of Participants With Clinically-Significant Change From Baseline in Neurological Examination Findings | Baseline up to 10 days after last dose of study intervention (approximately 5 weeks)

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of PF-07291177 | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 post-dose in each period
Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUClast) of PF-07291177 | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 post-dose in each period
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of PF-07291177 | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 post-dose in each period
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-07291177 | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 post-dose in each period
Plasma Half-Life (t1/2) of PF-07291177 | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 post-dose in each period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4741003